CLINICAL TRIAL: NCT06589622
Title: The Major Failures of Hall Technique Versus Atraumatic Restorative Technique in the Management of Carious Primary Molars: Randomized Clinical Trial
Brief Title: Major Failure Rate Assessment of Atraumatic Restorative Techniques Versus Hall Technique in the Management of Decayed Primary Molars in Children Aged 4-6 Years Old
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Norhan ahmed ibrahim ismail, principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ART vs Hall technique
Record Dates: First submitted 2024-09-06; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Decayed Primary Molars
Keywords: ART; Hall technique; decayed primary molars
MeSH Terms: interventions — Dental Atraumatic Restorative Treatment

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ART (Experimental): Atraumatic restorative technique
  Interventions: Procedure: Atraumatic Restorative Treatment
- Hall technique (Experimental): Stainless steel crown placement without tooth preparation
  Interventions: Procedure: Hall technique

INTERVENTIONS:
Procedure: Atraumatic Restorative Treatment — Caries excavation with hand instruments only and restoration with Glass ionomer filling
  Arms: ART
Procedure: Hall technique — Crown placement without tooth preparation
  Arms: Hall technique

SUMMARY:
This study is designed to compare major failure rate between ART ( excavation of caries with hand instruments and placing glass ionomer restoration without the use of rotary instruments) versus hall technique ( placing a stainless steel crown on the decayed primary molar without prepartion or caries removal)

ELIGIBILITY:
Inclusion Criteria

* Age: From 4 to 6 years.
* Cooperative children
* Children with no systemic disease, occlusal problems or bad habits.
* Primary molars with vital pulp.
* Class II Caries in primary molars within enamel/dentin.
* Molars in occlusion with the antagonist tooth/teeth.
* Teeth with no developmental anomalies.
* Absence of spontaneous pain and tenderness to percussion.
* Absence of any radiolucency in furcation and/or periradicular regions.
* No pathological and internal/external resorption.

Exclusion criteria:

* Presence of signs and symptoms of necrosis (Fistula, abscess, mobility or furcation involvement).
* Root caries.
* History of Spontaneous pain.

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 64 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Major failure | 1 year follow up
  Irreversible pulpitis, Dental abscess or fistula, Restoration loss, Tooth cannot be restored, Tooth fracture.

SECONDARY OUTCOMES:
Canine overbite | 3 months, 6 months and 1 year follow up
Postoperative pain and discomfort | Immediately postoperative
  Face pain scale-revised Its a self report measure of pain intenisty from 0 to 10 with 0 being least painful and 10 being most painful
Child anxiety | Intraoperative
  Venham anxiety rating scale is a scale from 0 to 5 assessing the anxiety of children in dental setting with 0 being most relaxed and smiling and 5 being most anxious and out of contact with the reality of the threat.
Child behavior | Intraoperative
  Venham behavior rating scale Its a scale from 0-5 with 0 being total cooperation and 5 being total uncooperation and physical restraint is required.

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: CSR